CLINICAL TRIAL: NCT07402252
Title: Effectiveness and Safety of a Type A Dissection Total Endovascular REconstruction System in Promoting Favorable Distal AOrtic ReModeling After Total Arch Replacement With Frozen Elephant Trunk for Type A Aortic Dissection: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Effectiveness and Safety of a Type A Dissection Total Endovascular Reconstruction System in Promoting Favorable Distal Aortic Remodeling
Acronym: REFORM-TAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jia Hu, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX2025001
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Residual Dissection After Repair for Type A Aortic Dissection
MeSH Terms: interventions — Surgical Procedures, Operative; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Standard medical therapy (e.g., blood pressure and heart rate control) plus endovascular repair with Study device following the Total Arch Replacement with Frozen Elephant Trunk for Stanford Type A Aortic Dissection.
  Interventions: Device: surgical treatment; Drug: Standard of Care (Investigator Choice)
- Control Group (Active Comparator): Standard medical therapy (e.g., blood pressure and heart rate control) without endovascular repair with Study device following the Total Arch Replacement with Frozen Elephant Trunk for Stanford Type A Aortic Dissection.
  Interventions: Drug: Standard of Care (Investigator Choice)

INTERVENTIONS:
Device: surgical treatment — Endovascular repair with study device following the Total Arch Replacement with Frozen Elephant Trunk for Stanford Type A Aortic Dissection.
  Arms: Study Group
Drug: Standard of Care (Investigator Choice) — Standard medical therapy (e.g., blood pressure and heart rate control)

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical study. A total of 198 eligible subjects will be enrolled and randomly assigned in a 1:1 ratio to either the Study Group or the Control Group. Subjects in the Study Group will receive surgical treatment using the study device (Type A Dissection Total Endovascular Reconstruction System) in addition to standard medical therapy following the Total Arch Replacement with Frozen Elephant Trunk. Subjects in the Control Group will continue standard medical therapy without surgical treatment using the study device following Total Arch Replacement with Frozen Elephant Trunk. Clinical follow-ups will be conducted at 30 days (±7 days), 6 months (±30 days), and 12 months (±30 days) post-enrollment to evaluate the effectiveness and safety of the study device.

After all subjects complete the 12-month (±30 days) follow-up, a statistical analysis will be performed and the results will be submitted for the study device registration application. Long-term follow-up will continue for 2-5 years post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Within 90 days of onset of Stanford Type A Aortic Dissection and 30 days post Total Arch Replacement with Frozen Elephant Trunk treatment (assessed via CTA at 30±7 days post open surgery):

   1. Presence of any intimal tear in the residual dissection of the thoracic aorta and the false lumen is not completely thrombosed.
   2. The intercostal arteries in the segment of the residual thoracic aortic dissection are primarily supplied by the false lumen (number of intercostal arteries supplied by false/mixed lumen > number supplied by true lumen; only intercostal arteries filled with contrast agent are considered).
   3. False lumen volume in the thoracic aorta distal to the frozen elephant trunk stent graft is >50% of the total aortic lumen volume.
3. Voluntarily participate in this study and provide signed informed consent.

Exclusion Criteria:

1. Presence of a proximal anastomotic leak at the frozen elephant trunk site post open surgery.
2. No left subclavian artery revascularization during the open surgery.
3. Presence of severe endoleak, or residual dissection expansion ≥55mm, or distal stent graft-induced new entry.
4. History of myocardial infarction, or stroke (with clear symptoms/signs and culprit lesion), or bowel ischemia within 1 month prior to the procedure.
5. Previous history of descending thoracic or abdominal aortic surgery.
6. Lack of suitable vascular access.
7. Known allergy to components of the study device (e.g., Nitinol) or contrast agent.
8. Renal insufficiency (creatinine >2.5 times the upper limit of normal) or requiring long-term regular dialysis.
9. Severe liver dysfunction (Child-Pugh Class C).
10. Active bleeding, coagulation disorders, thrombocytopenia (platelet count <50×109/L), or refusal of blood transfusion.
11. Uncontrolled severe infection and associated sepsis, shock, or multiple organ failure.
12. Life expectancy less than 12 months (due to conditions other than aortic dissection).
13. Known or suspected connective tissue degenerative disease, or family history of aortic dissection.
14. Pregnant or lactating women.
15. Concurrent participation in other drug or medical device clinical studies.
16. Subjects deemed unsuitable for participating the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in False Lumen Volume of the Distal Aortic Dissection at 12 months | 12 months (±30 days) post-enrollment
  Defined as the difference in the false lumen volume of the distal aortic dissection (distal to the frozen elephant trunk stent, including thrombosis portions) at baseline and 12 months (±30 days) post-enrollment among subjects in the Study group and Control group, respectively
The incidence of major adverse events (MAEs) within 30 days | 30 days (±7 days) after enrollment
  The percentage of subjects in the study or control group who experience any MAEs within 30 days (±7 days) after enrollment, relative to the total number of subjects in each group.

SECONDARY OUTCOMES:
Procedure Success Rate (%) (Immediate post-procedure) (Study Group only) | Immediately post procedure
  The percentage of subjects in the study group who achieved procedure success immediately after procedure out of the total number of subjects in the study group. Procedure success is defined as successful delivery and positioning of the system, accurate deployment of the stent, successful retrieval of the delivery system, no conversion to open surgical thoracotomy during the procedure, subject survival at the end of the procedure, and no Type I or III endoleak on angiography in the covered stent-graft segment.
Treatment Success Rate (%) (12 months) (Study Group only) | 12 months (±30 days) after enrollment
  The percentage of subjects in the study group who achieved treatment success at 12 months (±30 days) after enrollment out of the total number of subjects in the study group.
Change in True Lumen Volume of the Distal Aortic Dissection (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment.
  The difference in the volume change of the true lumen of distal aortic dissection (distal to the frozen elephant trunk stent, thoracic and abdominal segments) at baseline, 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) post-enrollment among subjects in the Study group and Control group, respectively.
Change in False Lumen Volume of the Distal Aortic Dissection (at 30 days, 6 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), and 2-5 years (±30 days) after enrollment
  The difference of change in the false lumen volume of distal aortic dissection (distal to the frozen elephant trunk stent, thoracic and abdominal segments, including thrombosis portions) at baseline, 30 days (±7 days), 6 months (±30 days), and 2-5 years (±30 days) post-enrollment among subjects in the Study group and Control group, respectively.
Change in Maximum Diameter of the Distal Aorta (True + False Lumen) (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment
  The difference in the maximum diameter change of the entire distal aorta (true lumen + false lumen, distal to the frozen elephant trunk stent, thoracic and abdominal segments) at baseline, 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) ost-enrollment among subjects in the Study group and Control group, respectively.
Thrombosis Status of the False Lumen in the Distal Aortic Dissection (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment
  The qualitative and/or quantitative assessment of thrombosis status in the false lumen of distal aortic dissection (aortic segment from the distal end of the frozen elephant trunk stent to the superior edge of the celiac trunk origin) for subjects in the study or control group at 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) post-enrollment, based on CTA imaging and aortic reconstruction models.
Rate of Secondary Intervention Related to the Distal Aortic Dissection (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment.
  The percentage of subjects in the study or control group who meet the indications for secondary intervention related to distal aortic dissection within 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) post-enrollment, relative to the total number of subjects in each group.
Survival Rate (6, 12 months, 2-5 years) | 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment
  The percentage of subjects in the study or control group with no all-cause death or aortic-related death at 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment, relative to the total number of subjects in each group.
Incidence of MAE (6, 12 months, 2-5 years) | 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment
  MAEs include any of the following aortic-related events: death, stroke, myocardial infarction, paraplegia/spinal cord ischemia, intestinal ischemia/necrosis requiring intervention, new-onset renal failure requiring replacement therapy, or respiratory failure requiring prolonged mechanical ventilation or reintubation.
Incidence of Paraplegia/Spinal Cord Ischemia (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment.
  The percentage of subjects in the study or control group who develop paraplegia or spinal cord ischemia within 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment, relative to the total number of subjects in each group.
Incidence of Acute Kidney Injury (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment.
  The percentage of subjects in the study or control group who develop acute kidney injury within 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment, relative to the total number of subjects in each group.
Incidence of Stroke (at 30 days, 6, 12 months, 2-5 years) | 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment
  The percentage of subjects in the study or control group who experienced a stroke within 30 days (±7 days), 6 months (±30 days), 12 months (±30 days), and 2-5 years (±30 days) after enrollment, relative to the total number of subjects in each group.
Incidence of Stent Migration (at 30 days, 6, 12 months) (Study Group only) | 30 days (±7 days), 6 months (±30 days), and 12 months (±30 days) after enrollment.
  The percentage of subjects in the study group with stent displacement within 30 days (±7 days), 6 months (±30 days), and 12 months (±30 days) after enrollment, relative to the total number of subjects in each group.
Incidence of AE/SAEs | Through study completion, an average of 5 year
  AE refers to any unfavorable medical event occurring during a clinical trial, whether or not related to the study device.
Incidence of Device Deficiencies (Study Group only) | Through study completion, an average of 5 year
  A device deficiency refers to any unreasonable risk that may endanger human health and safety during normal use of the medical device in a clinical trial, such as label errors, quality issues, malfunctions, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China